CLINICAL TRIAL: NCT06371118
Title: HPV Self-sampling for Women Who do Not Attend the Organized Cervical Cancer Screening Programme (HERSELF)
Brief Title: HPV Self-sampling for Women Who do Not Attend Cervical Cancer Screening Programme
Acronym: HERSELF
Status: Recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: Universidade do Porto (Other)
Collaborators: Unidade de Saúde Familiar de Garcia de Orta, Porto (Unknown); Unidade de Saúde Familiar da Prelada, Porto (Unknown); Unidade de Saúde Familiar de Cedofeita, Porto (Unknown); Instituto Portugues de Oncologia, Francisco Gentil, Porto (Other)
Responsible Party: Principal Investigator, Maria Margarida Martins Novais Teixeira, Medical Doctor, Instituto de Saude Publica da Universidade do Porto
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Diagnostic
Other Study IDs: PI 20210032
Record Dates: First submitted 2024-04-09; First posted 2024-04-17 (Actual); Last update posted 2024-05-14 (Actual); Status verified 2024-05

CONDITIONS: Papillomavirus Infections; Early Detection of Cancer; Cervix Cancer; Self-Examination
MeSH Terms: conditions — Papillomavirus Infections; Uterine Cervical Neoplasms; Self-Examination

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (3):
- Control group (Active Comparator): An invitation to attend a cervical cancer screening in a clinical setting will be sent by post to the woman's address.
  Interventions: Diagnostic Test: Standard of care - screening in a clinical setting
- Intervention 1 (directly mailed group) (Experimental): The HPV self-sampling test will be sent by post directly to the woman's address.
  Interventions: Device: Directly mailed self-sampling kit to collect a vaginal sample
- Intervention 2 (opt-in group) (Experimental): The HPV self-sampling test will be sent by post directly to the woman's address after a opt-in procedure.
  Interventions: Device: Mailed self-sampling kit to collect a vaginal sample after opt-in prodecure

INTERVENTIONS:
Device: Directly mailed self-sampling kit to collect a vaginal sample — The HPV self-sampling test will be sent by post directly to the woman's address. If the woman does not return the sample within 20 days, she will be sent a SMS reminder.
  The returned samples will be analysed. If high-risk HPV is present, women will be invited to be screened for cervical cancer in a clinical setting by their family doctors.
  Self-samples in which high-risk HPV is present will also be subjected to HPV DNA methylation test. If an abnormal HPV DNA methylation is detected and the woman has not attended the screening in a clinical setting yet, she will be informed by her family doctor that a new test has indicated the need to attend a medical appointment.
  Other Names: Evalyn Brush
  Arms: Intervention 1 (directly mailed group)
Device: Mailed self-sampling kit to collect a vaginal sample after opt-in prodecure — Women will initially receive an invitation letter in their home addresses to receive the self-sampling kit, as well as a pre-paid envelope to return the answer to this invitation. If the woman does not return the answer within 10 days, she will be sent a SMS reminder. Only those who respond affirmatively to the question will receive the self-sampling kit.
  The steps that follow will be the same as in intervention 1.
  Other Names: Evalyn Brush
  Arms: Intervention 2 (opt-in group)
Diagnostic Test: Standard of care - screening in a clinical setting — Corresponds to the standard of care. An invitation to attend the conventional cervical cancer screening (clinician-collected cervical sample for HPV test and reflex cytology) will be sent by post to the woman's address.
  Arms: Control group

SUMMARY:
This study aims to test the effectiveness and cost-effectiveness of two different strategies of home-delivered HPV self-sampling, in comparison to the standard of care strategy, to increase adherence to cervical cancer screening.

An experimental and population-based study will be implemented at three primary healthcare centers located in the Western Porto region: Cedofeita, Garcia de Orta, and Prelada. Eligible women will be randomized into a control group or an intervention group. The control group will correspond to the standard of care (invitation to screening in a clinical setting). The intervention group will be randomized into two subgroups: 1) a "directly mailed" group that will receive a self-sampling kit at their home addresses by post; 2) an "opt-in" group that will receive an invitation at home asking if they want to receive a self-sampling kit, with a pre-paid envelope to return the answer to this question. Women who answer "yes" will receive the self-sampling kit at their home addresses by post.

Self-sampling samples will be subjected to HPV genotyping. In parallel, high-risk HPV positive women will be called in by their family doctors to undergo screening in a clinical setting so that they can continue their clinical follow-up in the conventional pathway.

DETAILED DESCRIPTION:
The goal of this randomized clinical trial is to test the effectiveness and cost-effectiveness of two different strategies of home-delivered HPV self-sampling to increase the adherence to cervical cancer screening in women who are overdue for cervical cancer screening, in comparison to the standard of care strategy.

The main questions this study aims to answer are:

* To test the effectiveness of an invitation strategy to improve the adherence to cervical cancer screening based on directly home-delivered HPV self-sampling tests + automated reminders, in comparison to the standard of care invitation.
* To test the effectiveness of an invitation strategy to improve the adherence to cervical cancer screening based on home-delivered HPV self-sampling tests using opt-in procedures for ordering the kit + automated reminders, in comparison to the standard of care invitation.
* To compare the cost-effectiveness between a) standard of care; b) directly home-delivered HPV self-sampling tests + automated reminders; and c) home-delivered HPV self-sampling tests using opt-in procedures for ordering the kit + automated reminders.

Eligible women will be randomized (1:1) into a control group and an intervention group:

* Control group: corresponds to the standard of care, which is an invitation to cervical cancer screening in a clinical setting, through a written letter, printed and sent by the primary healthcare unit where the women are registered.
* Intervention group: Women allocated to this group will be randomized (1:1) into two subgroups, described briefly as follows:

  * Intervention 1 (half of the intervention group): HPV self-sampling test mailed directly to the women's home address (directly mailed group), complemented with a SMS reminder. If a woman returns the sample, HPV-type genotyping will be performed. If High-Risk HPV (HR-HPV) is detected, women will be informed of the result and invited to take cervical cancer screening in a clinical setting by their family doctors. Subsequent follow-up will take place according to Portuguese guidelines.
  * Intervention 2 (half of the intervention group): An invitation is mailed to the women´s home address, offering a self-sampling kit, to be ordered by returning a prepaid envelope with the answer "yes" (opt-in group). In the event of a positive response, an HPV self-sampling test is mailed to the women's home, complemented with a SMS reminder. If a woman returns the sample, HPV genotyping will be performed. If HR-HPV is detected, women will be informed of the result and invited to take cervical cancer screening in a clinical setting, performed by their family doctors. Subsequent follow-up will take place according to Portuguese guidelines.

In Interventions 1 and 2, when HR-HPV is detected in the self-sampling test, this sample will be subjected to HPV-DNA methylation testing. If increased HPV DNA methylation is detected and the woman has yet not attended the conventional screening invitation by her family doctor, she will be informed by her family doctor that a new test has indicated an increased risk for cervical cancer and the need to attend a medical appointment will be reinforced.

ELIGIBILITY:
Inclusion Criteria:

* Women aged between 26 and 60 years old;
* Women eligible for cervical cancer screening whose screening is at least 1 year overdue.

Exclusion Criteria:

* No mobile phone number available at the National Health Service database;
* Foreign mobile phone number;
* No address available at the National Health Service database;
* Foreign address.

Ages: 26 Years to 60 Years | Sex: Female | Healthy Volunteers: Yes
Age Groups: Adult
Gender Based: Yes — Women
Enrollment: 1000 (Estimated)
Dates: Start 2024-04-15 (Actual); Primary Completion 2024-09 (Estimated); Study Completion 2024-11 (Estimated)

PRIMARY OUTCOMES:
Adherence to conventional screening in control group | 45 and 90 days after the conventional screening appointment date
  Number of women in control group who adhered to conventional screening divided by the number of women assigned to control group
Adherence to HPV self-sampling in intervention 1 (directly mailed) group | 45 and 90 days after the day the self-sampling kit is sent
  Number of women who returned the self-sample in intervention 1 group divided by the number of women assigned to intervention 1 group
Adherence to HPV self-sampling in intervention 2 (opt-in) group | 45 and 90 days after the day the self-sampling kit is sent
  Number of women who returned the self-sample in intervention 2 group divided by the number of women assigned to intervention 2 group
Adherence proportion to HPV self-sampling in intervention 1 (directly mailed) group VS Adherence proportion to conventional screening in control group | 45 and 90 days after the day the self-sampling kit is sent or 45 and 90 days after the conventional screening appointment date, as appropriate
  The quotient of (Number of women in intervention 1 group who returned the self-sample divided by the women assigned to intervention 1 group) dividided by (Number of women in control group who adhered to conventional screening divided by the number of women assigned to control group).
Adherence proportion to HPV self-sampling in intervention 2 (opt-in) group VS Adherence proportion to conventional screening in control group | 45 and 90 days after the day the self-sampling kit is sent or 45 and 90 days after the conventional screening appointment date, as appropriate
  The quotient of (Number of women in intervention 2 group who returned the self-sample divided by the women assigned to intervention 2 group) dividided by (Number of women in control group who adhered to conventional screening divided by the number of women assigned to control group).

SECONDARY OUTCOMES:
Adherence to first follow-up step in control group | 45 and 90 days after the colposcopy appointment date
  Quotient of the number of women in control group who adhered to first follow-up step (in this case, colposcopy) divided by the number of women assigned to control group
Adherence to first follow-up step in intervention 1 (directly mailed) group | 45 and 90 days after the clinician-sampling appointment date
  Quotient of the number of women in intervention 1 group who adhered to first follow-up step (in this case, clinician-sampling) divided by the number of women assigned to intervention 1 group
Adherence to first follow-up step in intervention 2 (opt-in) group | 45 and 90 days after the clinician-sampling appointment date
  Quotient of the number of women in intervention 2 group who adhered to first follow-up step (in this case, clinician-sampling) divided by the number of women assigned to intervention 2 group
Adherence to first follow-up step in control group among women referred for follow-up | 45 and 90 days after the colposcopy appointment date
  Quotient of the number of women in control group who adhered to first follow-up step (in this case, colposcopy) divided by the number of women assigned to control group who were referred for follow-up (colposcopy) after an abnormal result in conventional screening
Adherence to first follow-up step in intervention 1 (directly mailed) group among women referred for folow-up | 45 and 90 days after the clinician-sampling appointment date
  Quotient of the number of women in intervention 1 group who adhered to first follow-up step (in this case, clinician-sampling) divided by the number of women assigned to intervention 1 group who were referred for follow-up (clinician-sampling) after an abnormal result in self-sampling
Adherence to first follow-up step in intervention 2 (opt-in) group among women referred for folow-up | 45 and 90 days after the clinician-sampling appointment date
  Quotient of the number of women in intervention 2 group who adhered to first follow-up step (in this case, clinician-sampling) divided by the number of women assigned to intervention 2 group who were referred for follow-up (clinician-sampling) after an abnormal result in self-sampling
Adherence to colposcopy in control group | 45 and 90 days after the colposcopy appointment date
  Quotient of the number of women in control group who adhered to colposcopy divided by the number of women assigned to control group
Adherence to colposcopy in intervention 1 (directly mailed) group | 45 and 90 days after the colposcopy appointment date
  Quotient of the number of women in intervention 1 group who adhered to colposcopy divided by the number of women assigned to intervention 1 group
Adherence to colposcopy in intervention 2 (opt-in) group | 45 and 90 days after the colposcopy appointment date
  Quotient of the number of women in intervention 2 group who adhered to colposcopy divided by the number of women assigned to intervention 2 group
Adherence to colposcopy in control group among women referred for colposcopy | 45 and 90 days after the colposcopy appointment date
  Quotient of the number of women in control group who adhered to colposcopy divided by the number of women assigned to control group who were referred for colposcopy after an abnormal result in conventional screening
Adherence to colposcopy in intervention 1 (directly mailed) group among women referred for colposcopy | 45 and 90 days after the colposcopy appointment date
  Quotient of the number of women in intervention 1 group who adhered to colposcopy divided by the number of women assigned to intervention 1 group who were referred for colposcopy after abnormal results in both self-sampling and clinician-sampling
Adherence to colposcopy in intervention 2 (opn-in) group among women referred for colposcopy | 45 and 90 days after the colposcopy appointment date
  Quotient of the number of women in intervention 2 group who adhered to colposcopy divided by the number of women assigned to intervention 2 group who were referred for colposcopy after abnormal results in both self-sampling and clinician-sampling
Timelapse (in days) between the shipment of self-sampling kit and the return of the sample, in intervention 1 (directly mailed) group | Follow-up will end at 90 days
  Adherence will be assessed using Kaplan-Meier survival analysis.
Timelapse (in days) between the invitation to receive a self-sampling kit and the return of the opt-in answer, in intervention 2 (opt-in) group | Follow-up will end at 90 days
  Adherence will be assessed using Kaplan-Meier survival analysis.
Timelapse (in days) between the shipment of self-sampling kit and the return of the sample, in intervention 2 (opt-in) group | Follow-up will end at 90 days
  Adherence will be assessed using Kaplan-Meier survival analysis.
Adherence proportion to first follow-up step in intervention 1 (directly mailed) group VS Adherence proportion to first follow-up step in control group | 45 and 90 days after the first follow-up step (clinician-sampling appointment date or colposcopy appointment date, as appropriate)
  The quotient of (Number of women in intervention 1 group who adhered to first follow-up step (in this case, clinician-sampling) divided by the number of women assigned to intervention 1 group) divided by (Number of women in control group who adhered to first follow-up step (in this case, colposcopy) divided by the number of women assigned to control group)
Adherence proportion to first follow-up step in intervention 2 (opt-in) group VS Adherence proportion to first follow-up step in control group | 45 and 90 days after the first follow-up step (clinician-sampling appointment date or colposcopy appointment date, as appropriate)
  The quotient of (Number of women in intervention 2 group who adhered to first follow-up step (in this case, clinician-sampling) divided by the number of women assigned to intervention 2 group) divided by (Number of women in control group who adhered to first follow-up step (in this case, colposcopy) divided by the number of women assigned to control group)
Adherence proportion to first follow-up step in intervention 1 (directly mailed) group among women referred for follow-up VS Adherence proportion to first follow-up step in control group among women referred for follow-up | 45 and 90 days after the first follow-up step (clinician-sampling appointment date or colposcopy appointment date, as appropriate)
  The quotient of (Number of women in intervention 1 group who adhered to first follow-up step (in this case, clinician-sampling) divided by the number of women assigned to intervention 1 group who were referred for follow-up (clinician-sampling) after an abnormal result in self-sampling) divided by (Number of women in control group who adhered to first follow-up step (in this case, colposcopy) divided by the number of women assigned to control group who were referred for follow-up (colposcopy) after an abnormal result in conventional screening)
Adherence proportion to first follow-up step in intervention 2 (opt-in) group among women referred for follow-up VS Adherence proportion to first follow-up step in control group among women referred for follow-up | 45 and 90 days after the first follow-up step (clinician-sampling appointment date or colposcopy appointment date, as appropriate)
  The quotient of (Number of women in intervention 2 group who adhered to first follow-up step (in this case, clinician-sampling) divided by the number of women assigned to intervention 2 group who were referred for follow-up (clinician-sampling) after an abnormal result in self-sampling) divided by (Number of women in control group who adhered to first follow-up step (in this case, colposcopy) divided by the number of women assigned to control group who were referred for follow-up (colposcopy) after an abnormal result in conventional screening)
Adherence proportion to colposcopy in intervention 1 (directly mailed) group VS Adherence proportion to colposcopy in control group | 45 and 90 days after the colposcopy appointment date
  The quotient of (Number of women in intervention 1 group who adhered to colposcopy divided by the number of women assigned to intervention 1 group) divided by (Number of women in control group who adhered to colposcopy divided by the number of women assigned to control group)
Adherence proportion to colposcopy in intervention 2 (opt-in) group VS Adherence proportion to colposcopy in control group | 45 and 90 days after the colposcopy appointment date
  The quotient of (Number of women in intervention 2 group who adhered to colposcopy divided by the number of women assigned to intervention 2 group) divided by (Number of women in control group who adhered to colposcopy divided by the number of women assigned to control group)
Adherence proportion to colposcopy in intervention 1 (directly mailed) group among women referred for colposcopy VS Adherence proportion to colposcopy in control group among women referred for colposcopy | 45 and 90 days after the colposcopy appointment date
  The quotient of (Number of women in intervention 1 group who adhered to colposcopy divided by the number of women assigned to intervention 1 group who were referred for colposcopy after an abnormal result in both self-sampling and clinician-sampling) divided by (Number of women in control group who adhered to colposcopy divided by the number of women assigned to control group who were referred for colposcopy after an abnormal result in conventional screening)
Adherence proportion to colposcopy in intervention 2 (opt-in) group among women referred for colposcopy VS Adherence proportion to colposcopy in control group among women referred for colposcopy | 45 and 90 days after the colposcopy appointment date
  The quotient of (Number of women in intervention 2 group who adhered to colposcopy divided by the number of women assigned to intervention 2 group who were referred for colposcopy after an abnormal result in both self-sampling and clinician-sampling) divided by (Number of women in control group who adhered to colposcopy divided by the number of women assigned to control group who were referred for colposcopy after an abnormal result in conventional screening)
Proportion of HR-HPV positivity in control group | 45 and 90 days after the conventional screening appointment date
  The quotient of the number of women in control group who tested positive for HR-HPV in conventional screening divided by the number of women assigned to control group
Proportion of HR-HPV positivity in intervention 1 (directly mailed) group | 45 and 90 days after the day the self-sampling kit is sent
  The quotient of the number of women in intervention 1 group who tested positive for HR-HPV in self-sampling divided by the number of women assigned to intervention 1 group
Proportion of HR-HPV positivity in intervention 2 (opt-in) group | 45 and 90 days after the day the self-sampling kit is sent
  The quotient of the number of women in intervention 2 group who tested positive for HR-HPV in self-sampling divided by the number of women assigned to intervention 2 group
Proportion of HR-HPV positivity in control group among women who adhered to conventional screening | 45 and 90 days after the conventional screening appointment date
  The quotient of the number of women in control group who tested positive for HR-HPV in conventional screening divided by the number of women assigned to control group who adhered to conventional screening
Proportion of HR-HPV positivity in intervention 1 (directly mailed) group among women who returned the self-sample | 45 and 90 days after the day the self-sampling kit is sent
  The quotient of the number of women in intervention 1 group who tested positive for HR-HPV in self-sampling divided by the number of women assigned to intervention 1 group who returned the self-sample
Proportion of HR-HPV positivity in intervention 2 (opt-in) group among women who returned the self-sample | 45 and 90 days after the day the self-sampling kit is sent
  The quotient of the number of women in intervention 2 group who tested positive for HR-HPV in self-sampling divided by the number of women assigned to intervention 2 group who returned the self-sample
Proportion of HR-HPV 16/18 positivity in control group | 45 and 90 days after the conventional screening appointment date
  The quotient of the number of women in control group who tested positive for HR-HPV 16/18 in conventional screening divided by the number of women assigned to control group
Proportion of HR-HPV 16/18 positivity in intervention 1 (directly mailed) group | 45 and 90 days after the day the self-sampling kit is sent
  The quotient of the number of women in intervention 1 group who tested positive for HR-HPV 16/18 in self-sampling divided by the number of women assigned to intervention 1 group
Proportion of HR-HPV 16/18 positivity in intervention 2 (opt-in) group | 45 and 90 days after the day the self-sampling kit is sent
  The quotient of the number of women in intervention 2 group who tested positive for HR-HPV 16/18 in self-sampling divided by the number of women assigned to intervention 2 group
Proportion of HR-HPV 16/18 positivity in control group among women who adhered to conventional screening | 45 and 90 days after the conventional screening appointment date
  The quotient of the number of women in control group who tested positive for HR-HPV 16/18 in conventional screening divided by the number of women assigned to control group who adhered to conventional screening
Proportion of HR-HPV 16/18 positivity in intervention 1 (directly mailed) group among women who returned the self-sample | 45 and 90 days after the day the self-sampling kit is sent
  The quotient of the number of women in intervention 1 group who tested positive for HR-HPV 16/18 in self-sampling divided by the number of women assigned to intervention 1 group who returned the self-sample
Proportion of HR-HPV 16/18 positivity in intervention 2 (opt-in) group among women who returned the self-sample | 45 and 90 days after the day the self-sampling kit is sent
  The quotient of the number of women in intervention 2 group who tested positive for HR-HPV 16/18 in self-sampling divided by the number of women assigned to intervention 2 group who returned the self-sample
Positive predictive value of self-sampling for the detection of HR-HPV, using clinician-sampling results as gold standard | 90 days after clinicial-sampling appointment date
  The quotient of the number of cases in which both self-sampling and clinician-sampling tested positive for HR-HPV divided by the number of cases in which self-sampling tested positive for HR-HPV, regardless of the clinician-sampling HR-HPV test result)
Sensitivity of HR-HPV testing and methylation analysis in self-samples, using biopsy results as gold standard | 90 days after the colposcopy appointment date
  The quotient of the number of self-samples with HR-HPV positive result, abnormal methylation result and ≥HSIL divided by the total number of self-samples with ≥HSIL
Specificity of HR-HPV testing and methylation analysis in self-samples, using biopsy results as gold standard | 90 days after the colposcopy appointment date
  The quotient of the number of self-samples with HR-HPV positive result, normal methylation result and ≤LSIL divided by the total number of self-samples with ≤LSIL
Positive likelihood ratio of HR-HPV testing and methylation analysis in self-samples, using biopsy results as gold standard | 90 days after the colposcopy appointment date
  The quotient of (Number of self-samples with HR-HPV positive result, abnormal methylation result and ≥HSIL divided by the total number of self-samples with ≥HSIL) divided by (The quotient of the number of self-samples with HR-HPV positive result, abnormal methylation result and ≤LSIL divided by the total number of self-samples with ≤LSIL)
Negative likelihood ratio of HR-HPV testing and methylation analysis in self-samples, using biopsy results as gold standard | 90 days after the colposcopy appointment date
  The quotient of (Number of self-samples with HR-HPV positive result, normal methylation result and ≥HSIL divided by the total number of self-samples with ≥HSIL) divided by (The quotient of the number of self-samples with HR-HPV positive result, normal methylation result and ≤LSIL divided by the total number of self-samples with ≤LSIL)
Accuracy of HR-HPV testing and methylation analysis in self-samples, using biopsy results as gold standard | 90 days after the colposcopy appointment date
  The quotient of (The sum of the number of self-samples with HR-HPV positive result, abnormal methylation result and ≥HSIL with the number of self-samples with HR-HPV positive result, normal methylation result and ≤LSIL) divided by the total number of self-samples with HR-HPV positive result, regardless of the methylation and biopsy results.
Sensitivity of HR-HPV non 16/18 testing and methylation analysis in self-samples, using biopsy results as gold standard | 90 days after the colposcopy appointment date
  The quotient of the number of self-samples with HR-HPV non 16/18 positive result, abnormal methylation result and ≥HSIL divided by the total number of self-samples with ≥HSIL
Specificity of HR-HPV non 16/18 testing and methylation analysis in self-samples, using biopsy results as gold standard | 90 days after the colposcopy appointment date
  The quotient of the number of self-samples with HR-HPV non 16/18 positive result, normal methylation result and ≤LSIL divided by the total number of self-samples with ≤LSIL
Positive likelihood ratio of HR-HPV non 16/18 testing and methylation analysis in self-samples, using biopsy results as gold standard | 90 days after the colposcopy appointment date
  The quotient of (Number of self-samples with HR-HPV non 16/18 positive result, abnormal methylation result and ≥HSIL divided by the total number of self-samples with ≥HSIL) divided by (The quotient of the number of self-samples with HR-HPV non 16/18 positive result, abnormal methylation result and ≤LSIL divided by the total number of self-samples with ≤LSIL)
Negative likelihood ratio of HR-HPV non 16/18 testing and methylation analysis in self-samples, using biopsy results as gold standard | 90 days after the colposcopy appointment date
  The quotient of (Number of self-samples with HR-HPV non 16/18 positive result, normal methylation result and ≥HSIL divided by the total number of self-samples with ≥HSIL) divided by (The quotient of the number of self-samples with HR-HPV non 16/18 positive result, normal methylation result and ≤LSIL divided by the total number of self-samples with ≤LSIL)
Accuracy of HR-HPV non 16/18 testing and methylation analysis in self-samples, using biopsy results as gold standard | 90 days after the colposcopy appointment date
  The quotient of (The sum of the number of self-samples with HR-HPV non 16/18 positive result, abnormal methylation result and ≥HSIL with the number of self-samples with HR-HPV non 16/18 positive result, normal methylation result and ≤LSIL) divided by the total number of self-samples with HR-HPV non 16/18 positive result, regardless of the methylation and biopsy results.
Sensitivity of HR-HPV 16/18 testing and methylation analysis in self-samples, using biopsy results as gold standard | 90 days after the colposcopy appointment date
  The quotient of the number of self-samples with HR-HPV 16/18 positive result, abnormal methylation result and ≥HSIL divided by the total number of self-samples with ≥HSIL
Specificity of HR-HPV 16/18 testing and methylation analysis in self-samples, using biopsy results as gold standard | 90 days after the colposcopy appointment date
  The quotient of the number of self-samples with HR-HPV 16/18 positive result, normal methylation result and ≤LSIL divided by the total number of self-samples with ≤LSIL
Positive likelihood ratio of HR-HPV 16/18 testing and methylation analysis in self-samples, using biopsy results as gold standard | 90 days after the colposcopy appointment date
  The quotient of (Number of self-samples with HR-HPV 16/18 positive result, abnormal methylation result and ≥HSIL divided by the total number of self-samples with ≥HSIL) divided by (The quotient of the number of self-samples with HR-HPV 16/18 positive result, abnormal methylation result and ≤LSIL divided by the total number of self-samples with ≤LSIL)
Negative likelihood ratio of HR-HPV 16/18 testing and methylation analysis in self-samples, using biopsy results as gold standard | 90 days after the colposcopy appointment date
  The quotient of (Number of self-samples with HR-HPV 16/18 positive result, normal methylation result and ≥HSIL divided by the total number of self-samples with ≥HSIL) divided by (The quotient of the number of self-samples with HR-HPV 16/18 positive result, normal methylation result and ≤LSIL divided by the total number of self-samples with ≤LSIL)
Accuracy of HR-HPV 16/18 testing and methylation analysis in self-samples, using biopsy results as gold standard | 90 days after the colposcopy appointment date
  The quotient of (The sum of the number of self-samples with HR-HPV 16/18 positive result, abnormal methylation result and ≥HSIL with the number of self-samples with HR-HPV positive result, normal methylation result and ≤LSIL) divided by the total number of self-samples with HR-HPV 16/18 positive result, regardless of the methylation and biopsy results.

CONTACTS AND LOCATIONS:
Overall Officials: Maria Margarida MN Teixeira, MD, Principal Investigator — Instituto de Saude Publica da Universidade do Porto; Nuno Lunet, PhD, Study Chair — Instituto de Saude Publica da Universidade do Porto
Locations (2):
- Portugal (2):
  - Unidade de Saúde Familiar Cedofeita, Porto
  - Unidade de Saúde Familiar Prelada, Porto

IPD SHARING:
Plan to Share IPD: No